CLINICAL TRIAL: NCT04701710
Title: A Randomized Trial - Intensive Treatment Based in Ivermectin and Iota-carrageenan as Prophylaxis for Covid-19 In Healthcare Agents
Brief Title: Prophylaxis Covid-19 in Healthcare Agents by Intensive Treatment With Ivermectin and Iota-carrageenan
Acronym: Ivercar-Tuc
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Maria de los Angeles Peral de Bruno (Other Government)
Responsible Party: Sponsor-Investigator, Maria de los Angeles Peral de Bruno, Ph.D in Biological Science, Ministry of Public Health, Argentina
Organization: Ministry of Public Health, Argentina (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 5076-410-CH2020
Record Dates: First submitted 2021-01-07; First posted 2021-01-08 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Covid19; SARS (Severe Acute Respiratory Syndrome)
Keywords: Ivermectin; Iota-Carrageenan; Prophylaxis Covid-19; Healthcare Agents
MeSH Terms: conditions — COVID-19; Severe Acute Respiratory Syndrome | interventions — Ivermectin; Carrageenan

STUDY DESIGN:
Intervention Model Description: Randomized controlled 1:1. Experimental Group and Control Group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group (Experimental): The EG received Ivermectin orally 2 drops of 6 mg = 12 mg every 7 days, and Iota-Carrageenan 6 sprays per day for 4 weeks.
  Standard biosecurity care
  Interventions: Drug: Ivermectin / Iota-Carrageenan
- Control Group (No Intervention): Standard biosecurity care

INTERVENTIONS:
Drug: Ivermectin / Iota-Carrageenan — The EG received Ivermectin orally 2 drops of 6 mg = 12 mg every 7 days, and Iota-Carrageenan 6 sprays per day for 4 weeks.
  Other Names: Standard biosecurity care
  Arms: Experimental Group

SUMMARY:
IMPORTANCE: The emergency of COVID-19 requires the implementation of urgent strategies to prevent the spread of the disease, mainly in health personnel, who are the most exposed and has the highest risk of becoming infected with the SARS-COV-2.

OBJECTIVE: To evaluate the protective effect of the combination Ivermectin - Iota- Carrageenan, intensive treatment with repeated administration in oral- and nasal-spray, respectively, as a prophylaxis treatment prior to exposure to SARS-CoV-2, in health personnel at Public Healthcare Centers.

PARTICIPANTS, DESIGN AND SETTING: Randomized controlled 1-1 clinical trial in Personal Health, n = 234. The subjects were divided into experimental (EG)and control groups (CG). The EG received Ivermectin orally 2 drops of 6 mg = 12 mg every 7 days, and Iota-Carrageenan 6 sprays per day for 4 weeks. All participants were evaluated by physical examination COVID-19 diagnosed with negative RT-PCR at the beginning, final, and follow-up of the protocol. Differences between the variables were determined using the Chi-square test. The proportion test almost contagious subject and the contagion risk (Odd Ratio) were calculated using software STATA. The level of statistical significance was reached when p-Value < 0.05.

DETAILED DESCRIPTION:
The subjects were divided into experimental (EG: n=117; 39.6 +/- 9.4 years old, 65F) and control groups (CG: n=117; 38.4 +/- 7.4 years old, 61F).

RESULT: The number of subjects who were diagnosed with COVID-19 in GE was lower, only 4 of 117 (3.4%) than subjects in CG: 25 of 117 (21.4%) (p-Value = 0.0001). Twenty patients had mild symptoms (n= 4 in EG, n= 16 in CG), the proportion test was p-Value = 0.001. Six subjects were moderate, and 3 with severe diagnostics, all them in CG. The probability (Odd Ratio) of becoming ill with COVID-19 was significantly lower in EG with values of 0.13 (CI = [0.03, 0.40]; p-Value = 0.0001), this value (<1) indicates a protective effect of the Ivermectin / Iota-Carrageenan in the EG. Logistic regression test demonstrated that prophylactic in EG is independent of the patient's preexisting variable comorbidity was 0.11, CI= [0.04, 0.33], and p-Value= 0.0001. On the other hand, this variable was 2.78 CI= [1.19, 6.48], p-Value = 0.018 in CG. Also, we found that when increase the age variable, also increases contagious risk for Covid-19 in all subjects 0,93 CI=[0.88, 0.98], p-Value= 0,0012.

CONCLUSION: The intensive preventive treatment (short-term) with Ivermectin / Iota - Carrageenan was able to reduce the number of health workers infected with COVID-19. This treatment had an additional effect in preventing the severity of the disease, since most of the patients who received the treatment were mild. We propose a new therapeutic alternative for prevention and short-term intervention scheme (intensive) that is of benefit of the health worker in this pandemic accelerated time. This treatment did not produce lack of adherence or adverse effects.

Trial Registration: CEI (in Spanish: Comité de Ética en Investigación de la Dirección de Investigación del SI.PRO.SA, in English: Research Ethics Committee /Health Research Directorate) file number 52/2020.

ELIGIBILITY:
Inclusion Criteria:

* Personnel who perform patient care and administrative tasks:

  * medical personnel,
  * nurses,
  * kinesiologists,
  * orderlies,
  * administrative,
  * cleaning personnel.

Exclusion Criteria:

* People under 18 years of age,
* Pregnant or actively breastfeeding women,
* Presenting symptoms related to COVID-19 disease,
* Concurrent autoimmune or chronic disease,
* Immunosuppression,
* Active infectious diseases,
* History of previous SARSCoV-2 infection confirmed by RT-PCR or rapid test.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2020-12-18 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Pearson's Chi-square and proportion test. | 4 week
  Number of subjects who were diagnosed with COVID-19 in EG and CG.

SECONDARY OUTCOMES:
Odd Ratio, probabilistic test | 4 week
  Contagion risk. Severity and progression of symptoms.
Logistic regression test | 4 week
  Prophylactic effect associated with patient's preexisting comorbidity.

CONTACTS AND LOCATIONS:
Overall Officials: Rossana E Chahla, MD, Ph.D., Principal Investigator — Ministry of Health, Tucuman, Argentina
Locations (1):
- SI.PRO.SA, Ministerio de Salud Pública, San Miguel de Tucumán, Argentina

IPD SHARING:
Plan to Share IPD: No
N/C

REFERENCES:
- [Background] Caly L, Druce JD, Catton MG, Jans DA, Wagstaff KM. The FDA-approved drug ivermectin inhibits the replication of SARS-CoV-2 in vitro. Antiviral Res. 2020 Jun;178:104787. doi: 10.1016/j.antiviral.2020.104787. Epub 2020 Apr 3. PMID 32251768